CLINICAL TRIAL: NCT05887141
Title: Self-compassion and Self-criticism: a Virtual Reality Intervention
Acronym: VirtuS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: PPO (Unknown); University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10036
Record Dates: First submitted 2023-05-01; First posted 2023-06-02 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Self-Criticism
Keywords: Virtual Reality; self-criticism; self-compassion; perspective change; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Two independent substudies, each with two arms. N=68 per substudy (N=136 total)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (no perspective change) (Other): The intervention (two role-plays), however without using a perspective change afterwards.
  Interventions: Behavioral: Double Standards; Behavioral: Self-criticism avatar
- Perspective change condition (Experimental): The intervention (two role-plays) with a perspective change after each role-play.
  Interventions: Behavioral: Double Standards; Behavioral: Self-criticism avatar

INTERVENTIONS:
Behavioral: Double Standards — We created a VR intervention based on the Cognitive Behavioral Therapy (CBT) technique 'double standards'. In the intervention the participants have to respond to a virtual character they imagine as their friend, who expresses similar self-criticism as they struggle with themselves. Two role-plays are played in Virtual Reality (either with or without perspective change after the role-plays). In the perspective change condition, the perspective is changed with the virtual friend (second person perspective).
Behavioral: Self-criticism avatar — We created a VR intervention called 'Self-criticism avatar' that has common ground with two-chair dialogue. Participants have to assertively respond to their inner critic who criticizes them using their own self-critical thoughts. After responding assertively (for example: 'Go away, I don't need you', 'Good is good enough'), the virtual character becomes weaker until they give up. Two role-plays are played in Virtual Reality (either with or without perspective change after the role-plays). In the perspective change condition, the perspective is changed with a bystander (third person perspective).

SUMMARY:
The purpose of this study is to investigate two independent Virtual Reality interventions for self-criticism and self-compassion and the use of perspective-change in these interventions.

DETAILED DESCRIPTION:
The current study will use two novel Virtual Reality (VR) exercises that will be investigated through two independent sub-studies. First of all, an exercise that uses the CBT (Cognitive Behavioral Therapy) technique called 'Double standards'. People with excessive self-criticism often set higher standards for themselves, which makes them more critical towards themselves. A way to distance from this, to enable a more nuanced reflection, is to ask the patient what they would say to a friend having those same negative thoughts about themselves. Doing this utilizing a role play in a realistic VR environment of which the avatar has the characteristics of a friend, the effect could be even stronger. Furthermore, VR offers the chance to switch perspectives, in which the participants receive their own compassionate comments from the perspective of the friend, and experience themselves as a good friend.

The second exercise, 'Self-criticism avatar', has common grounds with the (two-)chair exercises of schema therapy and the voice dialogue method in which a patient enters a dialogue between one's inner voices. In the VR exercise, the participant will be able to choose a virtual character with a voice that represents their own inner critic and that gives them their own self-criticism. By assertively and strictly speaking up to the inner critic, after which the virtual character becomes smaller and smaller until it backs down, the participant can experience a sense of control over their self-criticism, which leaves more room for self-compassion. A discussion with the inner critic enables a more nuanced image with more self-compassion. The switch in perspective after the role-play allows the participant to see himself/herself speaking assertively to the avatar, which can strengthen the increase in self-compassion and decrease in self-criticism.

Switching of perspectives is a relatively new technique within VR, that can be of added value to regular psychological therapies. Regular psychological therapies use switching of perspectives by switching roles in a physical role-play between a therapist and a patient or in a group. Furthermore, imaginative switches of perspective are used in, for example, schema therapy or imagery rescripting. Even though this can bring new insight into another perspective, it is not possible to replay the role play where the participant can see himself/herself from someone else's perspective. This is, however, possible through VR.

The current study will investigate the two beforementioned VR exercises using two independent sub-studies, to determine whether they contribute to self-compassion and if the switch in perspective is of added value. This will be done by comparing two conditions for each VR exercise; one with a switch in perspective and one without a switch in perspective. The study aims to answer the following research questions:

* Do the two VR-self compassion exercises have a positive effect on self-compassion (increase) and self-criticism (decrease)?
* Is the switch in perspective for the exercise 'Double standards of added value? In other words: is receiving one's own compassionate response of added value in addition to showing compassion to a vulnerable other.
* Is the switch in perspective for the exercise 'self-criticism avatar' of added value? In other words: is watching oneself in a strong and resilient manner of added value in addition to assertively speaking up to one's inner critic?

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a study
* Score above 20 (>20) on the subscale 'Inadequate self' of the FSCRS questionnaire

Exclusion Criteria:

* N/A

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Self-Criticism and Self-Compassion Scales (SCCS) - Change in Self-Criticism | Right before (Timepoint 1) and directly after (Timepoint 2) the +/- 60 minute intervention
  Levels of state self-criticism as measured by the SCCS. The questionnaire consists of five scenarios that could induce self-critical and/or self-compassionate reactions. For the self-criticism scale, participants indicate on a 7-point Likert scale (1= not at all to 7= highly) to what extent they would react towards themselves in a contemptuous, critical, and harsh manner (range 15-105, higher scores reflect more self-criticism).
Self-Criticism and Self-Compassion Scales (SCCS) - Change in Self-Compassion | Right before (Timepoint 1) and directly after (Timepoint 2) the +/- 60 minute intervention
  Levels of state self-compassion as measured by the SCCS. The questionnaire consists of five scenarios that could induce self-critical and/or self-compassionate reactions. For the self-compassion scale, participants indicate on a 7-point Likert scale (1= not at all to 7= highly) to what extent they would react towards themselves in a reassuring, soothing, and compassionate manner (range 15-105, higher scores reflect more self-compassion).

SECONDARY OUTCOMES:
Change in negative affect | Right before (Timepoint 1) and directly after (Timepoint 2) the +/- 60 minute intervention
  Visual Analogue Scales (VAS) measuring negative affect with three questions (range 0-100 for each question, higher scores reflect a higher negative affect)
Change in positive affect | Right before (Timepoint 1) and directly after (Timepoint 2) the +/- 60 minute intervention
  Visual Analogue Scales (VAS) measuring positive affect with three questions (range 0-100 for each questions, higher scores reflect a higher positive affect)
Change in self-compassion and self-esteem | Right before (Timepoint 1) and directly after (Timepoint 2) the +/- 60 minute intervention
  Visual Analogue Scales (VAS) measuring self-compassion and self-esteem with six questions (range 0-100 for each question, higher scores reflect higher self-compassion and self-esteem)

OTHER OUTCOMES:
Demographics | Screening
  Age, gender and whether they've received psychological treatment in past/present
Forms of Self-Criticizing/Attacking and Self-Reassuring Scale (FSCRS) | Screening
  Trait levels of self-compassion and self-criticism as measured by the FSCRS. This questionnaire consists of 22 questions divided over 3 scales: 'Inadequate Self scale' (range 0-36, where higher scores reflect more self-criticism), 'Hated self' (range 0-20, where higher scores reflect more excessive self-criticism) and 'Reassured Self' (range 0-32, where higher scores reflect more self-compassion). Each question is answered on a 5-point Likert Scale (0= not at all like me; 4= extremely like me).
Evaluation questions | Directly after the +/- 60 minute intervention (Timepoint 2)
  A questionnaire asking participants what they thought of the intervention, consisting of nine questions answered on a 7-point Likert scale (with 1= strongly disagree and 7= strongly agree).
Igroup Presence questionnaire (IPQ) | Directly after the +/- 60 minute intervention (Timepoint 2)
  A questionnaire measuring presence in VR. The IPQ consists of 14 items that measure 3 subscales ('Spatial Presence', 'Involvement' and 'Experienced Realism') and has 1 item that measures the general 'sense of being there'. Participants answer the questions on a 7-point Likert scale ranging from -3 to +3.
Schema Mode Inventory, short version (SMI) | Right before the +/- 60 minute intervention (Timepoint 1)
  A questionnaire measuring the presence of 14 different schema modes (based on schema therapy). The questionnaire consists of 118 questions which participants answer on a 6 point Likert-scale (1= never/rarely, 6= always).
Suicide Probability Scale - Suicide Ideation | Right before the +/- 60 minute intervention (Timepoint 1)
  A questionnaire that measures the probability of suicide. For our study, we only included questions that measure the Suicide Ideation scale of the questionnaire. This scale consists of 8 questions that are answered on a 4-point Likert scale (0=Never/rarely to 3= Almost always/always). The range for the subscale Suicide Ideation is 0-24, where higher scores reflect more suicide ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Elise van der Stouwe, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from Marit Hidding, upon reasonable request.

REFERENCES:
- [Derived] Hidding M, Veling W, Pijnenborg GHM, van der Stouwe ECD. Facing your inner critic: a randomized controlled trial investigating a virtual reality intervention with and without a perspective change for excessive self-criticism. J Behav Ther Exp Psychiatry. 2025 Dec;89:102053. doi: 10.1016/j.jbtep.2025.102053. Epub 2025 Jul 16. PMID 40714698